CLINICAL TRIAL: NCT06300944
Title: The Effect of Low-dose Ketamine on Postoperative Pain Relief and Sleep Quality in Patients Undergoing Laparoscopic Uterine Surgery
Brief Title: The Effect of Esketamine on Postoperative Pain Relief in Patients Undergoing Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Ran Gao-2023-12
Record Dates: First submitted 2024-02-23; First posted 2024-03-08 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Postoperative Pain
Keywords: Esketamine; Laparoscopic uterine surgery; postoperative pain and sleep quality
MeSH Terms: conditions — Pain, Postoperative; Sleep Initiation and Maintenance Disorders | interventions — Sodium Chloride; Esketamine; Analgesics

STUDY DESIGN:
Intervention Model Description: parallel assignment
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group C(Control Group) (Active Comparator): At the beginning of the operation, intravenous infusion of reifentanil 0.1~0.2 μg/kg·min, propofol 2~4mg/kg·h, rocuronium 0.3mg/kg·h intermittently, inhalation of 1%~2% sevoflurane were maintained, the fluctuation of blood pressure was not more than 20% of the basic level, and the heart rate was 50~100 times /min. Pump proper amount of normal saline.The postoperative PCIA regimen was Sufentanil 2ug/kg, ondansetron 16mg, diluted with appropriate normal saline, a total of 100ml
  Interventions: Drug: saline
- Group K(Esketamine Group) (Experimental): Intraoperatively, remifentanil 0.1-0.2 μg/kg·min, propofol 2-4 mg/kg·h, intermittent rocuronium 0.3 mg/kg·h, inhalation of 1%-2% sevoflurane were given by continuous intravenous infusion, to maintain blood pressure fluctuation within 20% of the baseline level and heart rate within 50-100 beats/min. Esketamine 0.2mg/kg·h was pumped at the beginning of the procedure.The postoperative PCIA regimen was Sufentanil 2ug/kg, ondanseetron 16mg, esketamine 0.75mg/kg, diluted with appropriate normal saline, a total of 100ml.
  Interventions: Drug: Esketamine

INTERVENTIONS:
Drug: saline — A maintenance dose of saline is 0.2mg/kg/h and postoperative PCIA regimen was Sufentanil 2ug/kg, ondansetron 16mg, diluted with appropriate normal saline, a total of 100ml
  Other Names: placebo
  Arms: Group C(Control Group)
Drug: Esketamine — A maintenance dose of esketamine is 0.2mg/kg/h and postoperative PCIA regimen was Sufentanil 2ug/kg, ondanseetron 16mg, esketamine 0.75mg/kg, diluted with appropriate normal saline, a total of 100ml
  Other Names: analgesic
  Arms: Group K(Esketamine Group)

SUMMARY:
The purpose of this study is to investigate whether continuous intraoperative infusion of esketamine combined with the addition of esketamine to postoperative PCIA can improve postoperative pain and sleep quality in patients undergoing laparoscopic uterine surgery under general anesthesia.

DETAILED DESCRIPTION:
Esketamine is the right isomer of ketamine, which is better than the original ketamine and has fewer side effects. In addition, for some gynecological hysterectomy patients who have poor sleep quality and anxiety after surgery, Esketamine also has the effect of treating depression. Due to the side effects of postoperative nausea, vomiting and hyperalgesia caused by excessive dosage of some opioids, this study will continue to inject small doses of esketamine during the operation to reduce the intraoperative dosage of opioids, and add esketamine to the postoperative PCIA for analgesia. To explore whether this method can reduce the incidence of moderate and severe postoperative pain in patients with laparoscopic uterine surgery under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Patient Undergoing laparoscopic uterine surgery under general anesthesia (total hysterectomy, myomectomy);
2. Patients gave the informed consent and signed the informed consent form.
3. The ASA is Ⅰ-Ⅱ

Exclusion Criteria:

1. Patients allergic to anesthetics, ropivacaine, and esketamine or with contraindications to use;
2. Patients with cognitive dysfunction or an inability to communicate;
3. Transfer to the ICU after surgery;
4. Patients with hyperthyroidism, tachyarrhythmia, or severe hypertension;
5. Unwilling to use PCIA or refuse to participate in this trial;
6. Patients with liver and kidney dysfunction

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Moderate to severe pain | 2 hours, 4 hours, 8 hours, 12 hours, 24 hours after surgery
  Pain severity was measured using The NRS((Numerical Rating Scale), The NRS>3 was considered moderate to severe pain.The NRS score at 2 hours, 4 hours, 8 hours, 12hours, 24hours after surgery was observed to determine whether intraoperative infusion of esketamine combined with perioperative analgesia regimen of esketamine in postoperative PCIA could reduce the incidence of postoperative moderate to severe pain in patients undergoing gynecological laparoscopic uterine surgeryesketamine to postoperative PCIA can reduce the incidence of postoperative moderate to severe pain in patients undergoing laparoscopic uterine surgery under general anesthesia
Incidence of adverse reactions including nausea, vomiting and dizziness | Within 48 hours after surgery
  Postoperative nausea, vomiting and dizziness is the subjective discomfort of dizziness, nausea, vomiting after the patient is awake, and the diagnosis can be made according to the clinical manifestations of the patient after surgery. Incidence of adverse reactions including nausea, vomiting and dizziness within 48 hours after surgery.
Sleep quality | the first and second night after surgery
  Sleep quality scores on the first and second night after surgery was assessed by AIS((Athens Insomnia Scale).The AIS<4 was classified as no sleep disorder, AIS of 4 to 6 is classified as suspicious insomnia, AIS>6 is classified as insomnia.

SECONDARY OUTCOMES:
Remifentanil dosage | During surgery
  The total amount of remifentanil used during surgery
Additional post-operative analgesics | Within 48 hours after surgery
  The total amount of additional analgesics used after surgery (oral versus intramuscular)
Postoperative exhaust time of patients | Within three days after surgery
  How long does the patient recover bowel motility after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China

IPD SHARING:
Plan to Share IPD: No